CLINICAL TRIAL: NCT00771693
Title: Effects of Insulin Treatment on Postprandial Platelet Activation in Patients With NIDDM: a Placebo-controlled Dose-response Study With Insulin Aspart (Novorapid®)
Brief Title: Effects of Insulin Treatment on Postprandial Platelet Activation in Patients With Non-insulin-dependent Diabetes Mellitus (NIDDM)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Paul Hjemdahl, Professor, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: EudraCT number 2006-007031-27
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Type 2 Diabetes Mellitus; Postprandial Hyperglycemia
Keywords: NIDDM; Platelet Activation; Postprandial hyperglycemia; insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Insulin Resistance | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Insulin aspart (Novorapid®) — a cross-over study with subcutaneous injection of insulin aspart 0.1U/kg, 0.2u/kg or placebo, before the meal, on 3 different occasions.
  Other Names: NovoRapid (Novo-Nordisk)

SUMMARY:
The postprandial phase in diabetic patients is characterized by a rapid increase in blood glucose levels, increase in platelet aggregation, LDL oxidation and over production of thrombin.

The aim of the study is to determine whether meal induced platelet activation is related to post-prandial hyperglycemia, and can be attenuated by good postprandial glucose control with rapidly acting insulin in patients with T2DM.

DETAILED DESCRIPTION:
Each patient is admitted in the fasting state, on 3 different occasions . Blood glucose levels are normalized using intravenous infusion of insulin aspart , to a blood glucose level of 6-7 mmol/l. 15 minutes after normalization ,and right before a standardized meal, the patient is given a subcutaneous injection of insulin aspart 0.1 U/kg, 0.2 U/kg or placebo. The order of injections in the cross over study is randomized and blinded to the patient and to the investigators. The patient eats the meal and is followed up for 90 minutes after completion of the meal.

Blood tests for platelet function and other parameters are taken at 3 main points: 1. before glucose normalization.

2. 15 minutes after glucose normalization, and right before the meal. 3. 90 minutes after the meal.

Platelet function is evaluated by flow cytometry in whole blood (P- Selectin expression, Fibrinogen binding,aggregate formation: platelet- leukocyte, platelet-platelet, platelet-monocyte). Agonists that are used for platelet activation in flow cytometry are the thromboxane analogue U46619, ADP, and a collagen peptide that activates GPVI. Platelet adhesion is measured by the IMPACT cone and platelet analyser.

ELIGIBILITY:
Inclusion Criteria:

* Type II Diabetes Mellitus.
* Antecubital forearm veins allowing technically good sampling for platelet studies.
* HbA1c 6-9 % (Mono-S method).
* Below 70 years

Exclusion Criteria:

* History of a cardiovascular disease; Ischemic heart disease, Stroke, Peripheral vascular disease.
* Acute or chronic renal or liver disease
* Contraindication to insulin treatment
* Treatment with Glitazones, Sulphonylurea, antiplatelet drugs,
* Thrombocytopenia <150 X109/l.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To evaluate if platelet activation following a carbohydrate rich meal is related to the post-prandial hyperglycemia, and thus can be attenuated by premeal insulin treatment in patients with T2DM. | 90 minutes after the meal
Co- primary platelet response variables: U46619 stimulated platelet P- selectin activation, platelet-leukocyte aggregation, platelet-platelet aggregates and platelet-monocyte aggregates. | After completion of the study in 20 patients

SECONDARY OUTCOMES:
To elucidate if short-term lowering of blood glucose by insulin infusion (pretreatment standardization of blood glucose) reduces platelet activity in patients with T2DM. | After completion of the glucose normalization (before the meal)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hjemdahl, MD, PhD, Principal Investigator — Department of Medicine, Clinical Pharmacology Unit, Karolinska institute, Stockhom, Sweden
Locations (1):
- Department of Medicine, Clinical pharmacology Unit, Karolinska University Hospital, Solna., Stockholm, Sweden

REFERENCES:
- [Derived] Spectre G, Ostenson CG, Li N, Hjemdahl P. Postprandial platelet activation is related to postprandial plasma insulin rather than glucose in patients with type 2 diabetes. Diabetes. 2012 Sep;61(9):2380-4. doi: 10.2337/db11-1806. Epub 2012 Jun 11. PMID 22688337